CLINICAL TRIAL: NCT06267053
Title: Investigation of the Relationship Between Vitamin B12, Folic Acid and 25 OH D Levels and Radiologic Stage in Knee Osteoarthritis
Brief Title: Relationship Between Vitamins and Radiologic Stage in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Filiz Yildiz Aydin, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2023/469
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: Vitamin B12; Folate; Vitamin D; Gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Radiography, Dental, Digital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous blood was taken to serum-separating tube from the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kellgren Lawrence Grade: Patients are divided into four groups based on Kellgren lawrence stage
  Interventions: Diagnostic Test: Direct digital radiography; Diagnostic Test: 25-OH Vitamin D; Diagnostic Test: Vitamin B12; Diagnostic Test: Folic acid

INTERVENTIONS:
Diagnostic Test: Direct digital radiography — All the participants had anterior posterior and lateral knee xray taken within 3 months of diagnosis
Diagnostic Test: 25-OH Vitamin D — All the participants had serum 25-OH Vitamin D levels measured from venous blood within 30 days of diagnosis
Diagnostic Test: Vitamin B12 — All the participants had serum Vitamin B12 levels measured from venous blood within 30 days of diagnosis
Diagnostic Test: Folic acid — All the participants had serum folic acid levels measured from venous blood within 30 days of diagnosis

SUMMARY:
The aim of this study is to investigate the relationship between folic acid, vitamin B12 and 25-OH vitamin D levels and radiographic staging in patients diagnosed with primary gonarthrosis.

DETAILED DESCRIPTION:
While in the past osteoarthritis (OA) was believed to be a degenerative disease of cartilage alone, recently, many factors such as trauma, mechanical strain, inflammation, biochemical reactions, and metabolic irregularities have been shown to be involved in its etiology. Until now there have been many studies done to investigate the relationship between serum 25-OH Vitamin D (25(OH)D) levels and knee OA however the relationship between folic acid, vitamin B12 and knee OA has been rarely studied. Therefore, the aim of this study is to investigate the relationship between folic acid, vitamin B12 and 25(OH)D levels and radiographic staging in patients diagnosed with primary gonarthrosis.

The files of patients who presented to Sadi Konuk Training and Research Hospital's outpatient clinic of Physical Medicine and Rehabilitation with knee pain between June and December 2023 and were diagnosed with gonarthrosis according to the American College of Rheumatology (ACR) classification criteria were retrospectively reviewed.

Either one way ANOVA or Kruskal Wallis H test was used to compare means determined based on the result of the Shapiro Wilk test. Bonferroni PostHoc was used to compare between groups. The statistical analysis was performed with Statistical Package for the Social Sciences (SPSS) version 21 (New York, USA) with significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults (Age: 50-80) with primary gonarthrosis
* Anterior-posterior and lateral knee direct digital radiography within 3 months of diagnosis
* Vitamin B12, folic acid and 25-OH Vitamin D within 1 months of diagnosis

Exclusion Criteria:

* History of inflammatory or rheumatologic disease
* History of lower extremity surgery
* Pregnancy
* Active malignancy
* Severe mental disability

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patiens over 50 years old who presented to Bakirkoy Dr. Sadi Konuk Training and Reserach hospital's outpatient clinic of Physical Medicine and Rehabilitation with knee pain and diagnosed with gonarthrosis according to American College of Rheumatology (ACR) criteria
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
25-OH Vitamin D (25(OH)D) and Kellgren Lawrence Grade | Baseline
  One way ANOVA was used to determine the relationship between 25(OH)D and radiographical grade.
Vitamin B12 and Kellgren Lawrence Grade | Baseline
  Kruskal Wallis H Test was used to determine the relationship between Vitamin B12 and radiographical grade.
Folic acid and Kellgren Lawrence Grade | Baseline
  Kruskal Wallis H Test was used to determine the relationship between Folic acid and radiographical grade.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz YILDIZ AYDIN, Principal Investigator — Bakirkoy Dr. Sadi Konuk Research and Training Hospital; Sibel CAGLAR, Study Chair — Bakirkoy Dr. Sadi Konuk Research and Training Hospital; Arda Can KASAP, Study Chair — Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mora JC, Przkora R, Cruz-Almeida Y. Knee osteoarthritis: pathophysiology and current treatment modalities. J Pain Res. 2018 Oct 5;11:2189-2196. doi: 10.2147/JPR.S154002. eCollection 2018. PMID 30323653
- [Background] Gao XR, Chen YS, Deng W. The effect of vitamin D supplementation on knee osteoarthritis: A meta-analysis of randomized controlled trials. Int J Surg. 2017 Oct;46:14-20. doi: 10.1016/j.ijsu.2017.08.010. Epub 2017 Aug 7. PMID 28797917
- [Background] Perry TA, Parkes MJ, Hodgson R, Felson DT, O'Neill TW, Arden NK. Effect of Vitamin D supplementation on synovial tissue volume and subchondral bone marrow lesion volume in symptomatic knee osteoarthritis. BMC Musculoskelet Disord. 2019 Feb 14;20(1):76. doi: 10.1186/s12891-019-2424-4. PMID 30764805
- [Background] Namutebi F, Kayima J, Kaddumukasa M. Vitamin D and its association with symptom severity in knee osteoarthritis: a cross sectional study at a national referral hospital in Uganda. BMC Rheumatol. 2021 Dec 27;5(1):56. doi: 10.1186/s41927-021-00228-w. PMID 34955099
- [Background] Askari A, Ariya M, Davoodi SH, Shahraki HR, Ehrampoosh E, Homayounfar R. Vitamin K and D Status in Patients with Knee Osteoarthritis: An Analytical Cross-sectional Study. Mediterr J Rheumatol. 2021 Dec 27;32(4):350-357. doi: 10.31138/mjr.32.4.350. eCollection 2021 Dec. PMID 35128328
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Vargas-Uricoechea H, Nogueira JP, Pinzon-Fernandez MV, Agredo-Delgado V, Vargas-Sierra HD. Population Status of Vitamin B12 Values in the General Population and in Individuals with Type 2 Diabetes, in Southwestern Colombia. Nutrients. 2023 May 18;15(10):2357. doi: 10.3390/nu15102357. PMID 37242240
- [Background] Singh G, Hamdan H, Singh V. Clinical utility of serum folate measurement in tertiary care patients: Argument for revising reference range for serum folate from 3.0 ng/mL to 13.0 ng/mL. Pract Lab Med. 2015 Mar 26;1:35-41. doi: 10.1016/j.plabm.2015.03.005. eCollection 2015 Apr 1. PMID 28932797
- [Background] Agostini D, Donati Zeppa S. Vitamin D, Diet and Musculoskeletal Health. Nutrients. 2023 Jun 27;15(13):2902. doi: 10.3390/nu15132902. PMID 37447228
- [Background] Malas FU, Kara M, Kaymak B, Akinci A, Ozcakar L. Ultrasonographic evaluation in symptomatic knee osteoarthritis: clinical and radiological correlation. Int J Rheum Dis. 2014 Jun;17(5):536-40. doi: 10.1111/1756-185X.12190. Epub 2013 Oct 29. PMID 24618242
- [Background] Malas FU, Kara M, Aktekin L, Ersoz M, Ozcakar L. Does vitamin D affect femoral cartilage thickness? An ultrasonographic study. Clin Rheumatol. 2014 Sep;33(9):1331-4. doi: 10.1007/s10067-013-2432-y. Epub 2013 Nov 13. PMID 24221506
- [Background] Edd SN, Omoumi P, Jolles BM, Favre J. Longitudinal Femoral Cartilage T2 Relaxation Time and Thickness Changes with Fast Sequential Radiographic Progression of Medial Knee Osteoarthritis-Data from the Osteoarthritis Initiative (OAI). J Clin Med. 2021 Mar 21;10(6):1294. doi: 10.3390/jcm10061294. PMID 33801000
- [Background] Mermerci Baskan B, Yurdakul FG, Aydin E, Sivas F, Bodur H. Effect of vitamin D levels on radiographic knee osteoarthritis and functional status. Turk J Phys Med Rehabil. 2017 Apr 4;64(1):1-7. doi: 10.5606/tftrd.2018.986. eCollection 2018 Mar. PMID 31453483
- [Background] Bevilacqua G, Laskou F, Clynes MA, Jameson KA, Boucher BJ, Noonan K, Cooper C, Dennison EM. Determinants of circulating 25-hydroxyvitamin D concentration and its association with musculoskeletal health in midlife: Findings from the Hertfordshire Cohort Study. Metabol Open. 2021 Oct 26;12:100143. doi: 10.1016/j.metop.2021.100143. eCollection 2021 Dec. PMID 34755103
- [Background] Elbashir M, Shubayr N, Alghathami A, Ali S, Alyami A, Alumairi N, Abdelrazig A, Omer AM, Elbasheer O. Investigation of Vitamin D Status, Age, and Body Mass Index as Determinants of Knee Osteoarthritis Severity Using the Kellgren-Lawrence Grading System in a Saudi Arabian Cohort: A Cross-Sectional Study. Cureus. 2023 Oct 23;15(10):e47523. doi: 10.7759/cureus.47523. eCollection 2023 Oct. PMID 38021605
- [Background] Blom AB, van Lent PL, Holthuysen AE, van der Kraan PM, Roth J, van Rooijen N, van den Berg WB. Synovial lining macrophages mediate osteophyte formation during experimental osteoarthritis. Osteoarthritis Cartilage. 2004 Aug;12(8):627-35. doi: 10.1016/j.joca.2004.03.003. PMID 15262242
- [Background] de Visser HM, Korthagen NM, Muller C, Ramakers RM, Krijger GC, Lafeber FPJG, Beekman FJ, Mastbergen SC, Weinans H. Imaging of Folate Receptor Expressing Macrophages in the Rat Groove Model of Osteoarthritis: Using a New DOTA-Folate Conjugate. Cartilage. 2018 Apr;9(2):183-191. doi: 10.1177/1947603517738073. Epub 2017 Nov 3. PMID 29096521
- [Background] Xu H, Shin MH, Kang JH, Choi SE, Park DJ, Kweon SS, Lee YH, Kim HY, Lee JK, Lee SS. Folate deficiency is associated with increased radiographic severity of osteoarthritis in knee joints but not in hand joints. Clin Exp Rheumatol. 2023 May;41(5):1149-1154. doi: 10.55563/clinexprheumatol/69k9xr. Epub 2022 Oct 12. PMID 36226605
- [Background] Hong H, Chen L, Zhong Y, Yang Z, Li W, Song C, Leng H. Associations of Homocysteine, Folate, and Vitamin B12 with Osteoarthritis: A Mendelian Randomization Study. Nutrients. 2023 Mar 28;15(7):1636. doi: 10.3390/nu15071636. PMID 37049476
- [Background] Thomson A, Hilkens CMU. Synovial Macrophages in Osteoarthritis: The Key to Understanding Pathogenesis? Front Immunol. 2021 Jun 15;12:678757. doi: 10.3389/fimmu.2021.678757. eCollection 2021. PMID 34211470